CLINICAL TRIAL: NCT00002354
Title: One Year Study in HIV-1 Seropositive, AZT-Experienced Patients to Evaluate the Safety and Efficacy of MK-639 Administered Concomitantly With Stavudine (d4T)
Brief Title: A Study of Indinavir Sulfate Given Together With Stavudine to HIV-Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 246D; 37
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-01

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Stavudine; HIV Protease Inhibitors; Indinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Indinavir; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give indinavir sulfate plus stavudine to HIV-infected patients who have already been treated with zidovudine.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis with aerosolized pentamidine, topical antifungals, TMP / SMX, dapsone, or isoniazid.

Patients must have:

* HIV infection.
* CD4 count 50 - 500 cells/mm3.
* Prior AZT use for more than 6 months OR documented intolerance to AZT with more than 6 months use of another anti-HIV therapy other than d4T or any protease inhibitor.
* No active opportunistic infection or visceral Kaposi's sarcoma.

NOTE:

* Patients with hemophilia may be enrolled at discretion of investigator.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Symptomatic neuropathy.
* Acute hepatitis.

Concurrent Medication:

Excluded:

* Antiretrovirals other than specified in protocol.
* Chronic therapy for an active opportunistic infection.
* Immunosuppressive therapy.

Prior Medication:

Excluded:

* Any prior protease inhibitor or d4T.
* Any nucleoside analogs within 2 weeks prior to study entry.
* Investigational agents or immunomodulators within 30 days prior to study entry.

Required:

* More than 6 months of prior AZT unless intolerant, in which case more than 6 months of another anti-HIV therapy (other than protease inhibitors or d4T).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 540

CONTACTS AND LOCATIONS:
Locations (1):
- Merck & Co Inc, Whitehouse Station, New Jersey, United States